CLINICAL TRIAL: NCT00440414
Title: A Multicenter Randomized Phase III Study of Pemetrexed Versus Erlotinib in Patients With Pretreated Advanced Non-Small-Cell Lung Cancer (NSCLC)
Brief Title: Trial of Pemetrexed Versus Erlotinib in Pretreated Patients With Non Small Cell Lung Cancer (NSCLC)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hellenic Oncology Research Group (Other)
Collaborators: University Hospital of Crete (Other)
Responsible Party: L.Vamvakas, Hellenic Oncology Research Group
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT/06.05
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Last update posted 2010-08-19 (Estimated); Status verified 2010-08

CONDITIONS: Non Small Cell Lung Cancer
Keywords: Cancer; Non-small-cell lung cancer; Chemotherapy; Pemetrexed; Erlotinib
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Neoplasms | interventions — Erlotinib Hydrochloride; Pemetrexed

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): Alimta
  Interventions: Drug: Pemetrexed (Alimta)
- 2 (Experimental): Tarceva
  Interventions: Drug: Erlotinib (Tarceva)

INTERVENTIONS:
Drug: Erlotinib (Tarceva) — Erlotinib at the dose of 150 mg orally once a day continually until progression
  Other Names: Tarceva
  Arms: 2
Drug: Pemetrexed (Alimta) — Pemetrexed at the dose of 500mg/m2 IV infusion every 3 weeks for 6 consecutive cycles
  Other Names: Alimta
  Arms: 1

SUMMARY:
The second-line treatment in advanced NSCLC has been currently proved effective in prolonging overall survival and improving quality of life. Both pemetrexed and erlotinib have been approved for second-line treatment of NSCLC . Erlotinib is a valuable option for the treatment of advanced NSCLC, especially for elderly patients, due to convenience of administration and safety profile. The role of comprehensive geriatric assessment in treatment efficacy and tolerance is an area of investigation.

DETAILED DESCRIPTION:
This trial will compare the efficacy of pemetrexed versus erlotinib in pretreated patients with advanced NSCLC.

ELIGIBILITY:
Inclusion Criteria:

* Histologically- or cytologically- confirmed Non-Small-Cell Lung Cancer adenocarcinoma
* Stage IIIB/IV
* Failure to prior chemotherapy
* Presence of two-dimensional measurable disease. The measurable disease should not have been irradiated
* Absence or irradiated and stable central nervous system metastatic disease.
* Life expectancy of more than 3 months
* Tissue sample desired for genomic study
* Age ≥ 18 years
* Performance status (WHO) < 3
* For patients > 65 years old: "non-frail" according to comprehensive geriatric assessment
* Adequate bone marrow function (absolute neutrophil count > 1000/mm^3, platelet count > 100000/mm^3, hemoglobin > 9gr/mm^3)
* Adequate liver (bilirubin < 1.5 times upper limit of normal and SGOT/SGPT < 2 times upper limit of normal) and renal function (creatinine < 2mg/dl)
* Presence of a reliable care giver for patients > 65 years old
* Informed consent.

Exclusion Criteria:

* Psychiatric illness or social situation that would preclude study compliance
* Other concurrent uncontrolled illness
* Other invasive malignancy within the past 5 years except nonmelanoma skin cancer

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2006-04; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Time to Tumor Progression | 1 year TTP

SECONDARY OUTCOMES:
Overall response rate | Objective responses confirmed by CT or MRI (on 3rd and 6th cycle)
Overall survival between the two treatment arms | 1 year OS
Quality of life assessment | Assessment every two cycles
Toxicity profile between the two treatment arms | Toxicity assessment on each chemotherapy cycles

CONTACTS AND LOCATIONS:
Overall Officials: Lampros Vamvakas, MD, Principal Investigator — University Hospital of Crete; Athanasios Karampeazis, MD, Principal Investigator — University Hospital of Crete
Locations (9):
- Greece (9):
  - University General Hospital of Alexandroupolis, Dep of Medical Oncology, Alexandroupoli
  - 401 Military Hospital, Medical Oncology Unit, Athens
  - Air Forces Military Hospital, Dep of Medical Oncology, Athens
  - IASO General Hospital of Athens, 1st Department of Medical Oncology, Athens
  - Laikon General Hospital, Medical Oncology Unit, Propedeutic Dep of Internal Medicine, Athens
  - Sismanogleio General Hospital, 1st, 2nd Department of Pulmonary Diseases, Athens
  - Sotiria General Hospital, 1st, 3rd, 8th Dep of Pulmonary Diseases, Athens
  - Metaxa's Anticancer Hospital of Piraeus,1st Dep of Medical Oncology, Piraeus
  - Theagenion Anticancer Hospital of Thessaloniki, Thessaloniki